CLINICAL TRIAL: NCT06164002
Title: Application of Artificial Intelligence in the Prediction of Clinical Performance, Marginal Fit and Fracture Resistance of Vertical Versus Horizontal Margin Designs Fabricated With Two Ceramic Materials
Brief Title: A I in the Prediction of Clinical Performance, Marginal Fit and Fracture Resistance of Vertical Versus Horizontal Margin Designs Fabricated With 2 Ceramic Materials
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Walaa Tarek Mohamed, assisstant lecturer, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: P-CR-23-04
Record Dates: First submitted 2023-08-16; First posted 2023-12-11 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Artificial Intelligence
MeSH Terms: interventions — Artificial Intelligence; Models, Biological

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group (I) (Experimental): Patients will be prepared with vertical "feather edge" margin design.
  Interventions: Other: change in restoration material and margin design.
- Group (II) (Experimental): Patients will be prepared with horizontal "shoulder" margin design.
  Interventions: Other: change in restoration material and margin design.
- Subgroup (A) (Experimental): Patients will receive zirconia ceramic crowns
  Interventions: Other: change in restoration material and margin design.
- Subgroup (B) (Experimental): Patients will receive hybrid ceramic crowns.
  Interventions: Other: change in restoration material and margin design.

INTERVENTIONS:
Other: change in restoration material and margin design. — comparing two different materials and two different designs. use artificial intelligence in the prediction of follow up results
  Other Names: Predicting the follow up results using the new (artificial intelligence "AI") model

SUMMARY:
The present study will be performed to evaluate application of artificial intelligence in the prediction of clinical performance, marginal fit and fracture resistance of vertical "feather-edge" versus horizontal "shoulder" margin designs fabricated with two ceramic materials (zirconia and hybrid ceramic)

DETAILED DESCRIPTION:
The objective of the present study is to characterize two different margin designs (vertical "feather-edge" and horizontal "shoulder") with two different ceramic materials (zirconia and hybrid ceramic) in terms of clinical performance, marginal fit and fracture resistance.

Primary outcome:

Predicting the follow up results using the new (artificial intelligence "AI") model for vertical "feather-edge" versus horizontal "shoulder" margin designs fabricated with two ceramic materials (zirconia and hybrid ceramic) that saves the clinical evaluation period, hence saves the expenses of the dental clinic.

Secondary outcome:

Evaluating the clinical performance, marginal fit and fracture resistance of vertical "feather-edge" versus horizontal "shoulder" margin designs fabricated with two ceramic materials (zirconia and hybrid ceramic).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range of patients should be 20-50 years old, able to read and sign the informed consent document. 2. Patient with posterior molars indicated for full coverage restorations. 3. Patient should be able to physically and psychologically tolerate conventional restorative procedures. 4. Patients who are willing to return for follow-up examination and evaluation. 5. Indicated molar should have adequate tooth preparation length to ensure proper retention and resistance form. 6. Patient with sound contralateral or adjacent tooth to the selected tooth requiring full coverage restoration.

Exclusion Criteria:

1. Patient in the growth stage with partially erupted teeth.
2. Patient with poor oral hygiene and motivation.
3. Pregnant women.
4. Patient with psychiatric problems or unrealistic expectations.
5. Patients with no opposing occluding dentition in the area intended for restoration.
6. Patients with parafunctional habits. -

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Artificial intelligence application assessment, laboratory marginal fit and fracture resistance | 6 months
  Predicting the follow up results using the new (artificial intelligence "AI") model for vertical "feather-edge" versus horizontal "shoulder" margin designs fabricated with two ceramic materials (zirconia and hybrid ceramic) that saves the clinical evaluation period, hence saves the expenses of the dental clinic.

SECONDARY OUTCOMES:
In-Vitro Study preparations. | 6 months
  Marginal Adaptation "feather-edge" versus horizontal "shoulder" margin designs fabricated with two ceramic materials (zirconia and hybrid ceramic).
In-Vitro Study | 6 months
  Fracture Resistance
In-Vivo Study | Baseline,3 months,6 months
  Clinical Examination

CONTACTS AND LOCATIONS:
Locations (1):
- Walaa Tarek El Hefnawy, Cairo, Al-Azhar University, Egypt

IPD SHARING:
Plan to Share IPD: No